CLINICAL TRIAL: NCT02375386
Title: CENTRAL MECHANISMS OF BODY BASED INTERVENTION FOR MUSCULOSKELETAL LOW BACK PAIN: Feasibility Assessment of Neurophysiological Measurement in Veterans With Low Back Pain
Brief Title: Feasibility Assessment of Neurophysiological Measurement in Veterans With LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201300827-N; 3R01AT006334-02S1 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Therapeutic Touch; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal manipulation (Experimental): Participants will receive a lumbar SMT technique previously described in the literature and commonly utilized for the treatment of low back pain . The SMT will be performed four times (two times on each side) in a 5-minute period. In addition, the following will be performed: Functional MRI (fMRI), Behavioral: Pain Sensitivity Testing, Questionnaires,Behavioral: Physical Impairment.
  Interventions: Procedure: Spinal manipulation; Procedure: fMRI; Behavioral: Pain Sensitivity Testing; Other: Questionnaires; Behavioral: Physical Impairment
- Therapeutic touch (Sham Comparator): Participants in this group will lie prone. The therapist will place both hands in contact with the participants' pelvis across the top of the posterior aspect of the sacrum and ilia and apply a downward force to keep the pelvis in contact with the table. This group accounts for effects of time and personal contact. The amount of "hands-on" contact will be equivalent between groups. Both groups will be given the same verbal instructions regarding the techniques performed. In addition, the following will be performed: Functional MRI (fMRI), Behavioral: Pain Sensitivity Testing, Questionnaires,Behavioral: Physical Impairment.
  Interventions: Procedure: Therapeutic touch; Procedure: fMRI; Behavioral: Pain Sensitivity Testing; Other: Questionnaires; Behavioral: Physical Impairment

INTERVENTIONS:
Procedure: Spinal manipulation — Participants will receive a lumbar SMT technique previously described in the literature and commonly utilized for the treatment of low back pain . The SMT will be performed four times (two times on each side) in a 5-minute period. In addition, the following will be performed: Functional MRI, Behavioral: Pain Sensitivity Testing, Questionnaires,Behavioral: Physical Impairment.
  Arms: Spinal manipulation
Procedure: Therapeutic touch — Participants in this group will lie prone. The therapist will place both hands in contact with the participants' pelvis across the top of the posterior aspect of the sacrum and ilia and apply a downward force to keep the pelvis in contact with the table. This group accounts for effects of time and personal contact. The amount of "hands-on" contact will be equivalent between groups. Both groups will be given the same verbal instructions regarding the techniques performed. In addition, the following will be performed: Functional MRI, Behavioral: Pain Sensitivity Testing, Questionnaires,Behavioral: Physical Impairment.
  Arms: Therapeutic touch
Procedure: fMRI — Both groups will receive an fMRI.
  Other Names: Functional MRI
Behavioral: Pain Sensitivity Testing — Both groups will receive an Pain Sensitivity Testing
Other: Questionnaires — Both groups will receive Questionnaires
Behavioral: Physical Impairment — Both groups will receive testing on physical impairment.

SUMMARY:
This is study testing the feasibility of collecting neurophysiological measures of outcome related to body-based interventions for low back pain. The investigators will collect fMRI and psychophysical data about pain sensitivity before and after the interventions. Participants will be randomly assigned to either spinal manipulation or therapeutic touch groups. Participants will attend two practice sessions prior to the first data collection. There will be two follow-up assessments.

DETAILED DESCRIPTION:
Participants will be enrolled from VA pain clinical at the North Florida/South George VA Medical Center.

The investigators will collect functional magnetic resonance imaging data of resting state and pain-related events (i.i. during thermal pain sensitivity testing, as well as psychophysical data to determine pain sensitivity. Pain sensitivity will be measured using thermal and mechanical stimuli. These data will be collected before and after the interventions, in addition to two follow-up sessions after intervention.

In addition, clinical measures of pain intensity in the low back, as well as trunk range of motion and strength will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* complaints of current back pain that they rate at least 40 on a 101-point numeric rating scale
* Participants must able to understand written and spoken English

Exclusion Criteria:

* currently receiving treatment for LBP or have received SMT for LBP in the past year
* Quebec Task Force on Spinal Disorders (QTFSD) to identify patients with pre-existing nerve root compression, spinal stenosis, or post-surgery
* any chronic medical conditions that may affect pain perception (e.g., diabetes, high blood pressure, fibromyalgia, headaches)
* any contraindication to MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
fMRI during testing of pain changes from approximately Day 3 and Day 5 | Change from approximately Day 3 and Day 5
fMRI during quite rest changes from approximately Day 3 and Day 5 | Change from approximately Day 3 and Day 5
Pain Sensitivity Testing changes from Day 3, Day 4 and Day 5 | Change from Day 3, Day 4 and Day 5
  This measure thermal threshold and tolerance using continuous heat stimulus delivered to the participants' dominant arm. The stimulus will start at 35°C and will be increased at a rate of 0.5°C with participants terminating the stimulus when the temperature reached pain threshold ("when the sensation first transitions from heat to pain") and tolerance ("when the sensation becomes so strong you want to remove it from your skin"). Threshold and tolerance measures will also be collected using mechanical pressure applied using a Fischer Dolorimeter. During Dolorimeter testing, force is slowly increased until the subject indicates that the sensation changes from pressure to pain.

SECONDARY OUTCOMES:
Pain Intensity | Change from Day 3, Day 4 and Day 5
  Pain visual analog scale is a 10cm long line. The line is anchored at one end with 'none' or 'not bad at all' and at the other with 'worst imaginable.' Participants are asked to rate their pain at rest by placing a mark along the 10cm line. Participants will also rate pain during active trunk range of motion using the same scale.
McGill Pain Questionnaire-2 | Change from Day 3, Day 4 and Day 5
  This is 22-item questionnaire that asks participants to describe the intensity of varies qualities of the pain that he or she is experiencing; for example, throbbing or itching.
Physical Impairment | Change from Day 3, Day 4 and Day 5
  A physical impairment scale consists of 7 different examination procedures that assess lumbar and hip range of motion, muscle performance of trunk musculature, and response to palpation. Scores is 0 - 8, Range is 0 is no impairment and 8 is completely impaired.
Oswestry Disability Questionnaire (ODQ) | Change from Day 3, Day 4 and Day 5
  The ODQ has a range of 0 (no disability due to back pain) to 100 (completely disabled due to back pain), so higher scores indicate higher disability from LBP.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Bishop, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No